CLINICAL TRIAL: NCT01577173
Title: A Phase II, Open-Label, Randomized Study of MEDH7945A Versus Cetuximab in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck Who Have Progressed During or Following Platinum-based Chemotherapy
Brief Title: A Study of MEHD7945A Versus Cetuximab in Patients With Recurrent/Metastatic Squamous Cell Carcinoma of The Head And Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28076; 2011-005539-22 (EudraCT Number)
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — MEHD7945A; Cetuximab

ARMS (2):
- A: MEHD7945A (Experimental)
  Interventions: Drug: MEHD7945A
- B: Cetuximab (Active Comparator)
  Interventions: Drug: cetuximab

INTERVENTIONS:
Drug: MEHD7945A — 1100 mg iv every 2 weeks
  Arms: A: MEHD7945A
Drug: cetuximab — 400 mg/m2 iv loading dose, followed by 250 mg/m2 weekly
  Arms: B: Cetuximab

SUMMARY:
This phase II, open-label, randomized study will evaluate the efficacy and safety of MEHD7945A versus cetuximab in patients with recurrent/metastatic squamous cell carcinoma of the head and neck who have progressed during or following platinum-based chemotherapy. Patients will be randomized to receive either MEHD7945A 1100 mg intravenously (iv) every 2 weeks or cetuximab 400 mg/m2 iv loading dose followed by 250 mg/m2 iv weekly. Patients treated with cetuximab (Arm B) may cross-over to MEHD7945A (Arm A) upon central confirmation of progressive disease and upon meeting eligibility criteria. Anticipated time on study treatment is until disease progression or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically confirmed Stage III or IV recurrent/metastatic squamous cell carcinoma of the head and neck (R/M SCCHN)
* Progressive disease on or after first-line platinum-based chemotherapy regimen for R/M SCCHN (maximum of 6 cycles)
* No more than one platinum-based chemotherapy regimen for R/M SCCHN is allowed
* Prior platinum-based treatment as definitive chemo/radiotherapy for locally advanced disease is allowed if completed/terminated >/= 6 months before the platinum-based regimen for R/M SCCHN
* Consent to provide archival tumor tissue for biomarker testing
* Measurable disease per RECIST v1.1
* ECOG performance status of 0, 1 or 2
* Adequate hematologic, renal and liver function

Exclusion Criteria:

* Nasopharyngeal cancer
* Prior treatment with an investigational or approved agent for the purpose of inhibiting HER family members
* This includes but is not limited to cetuximab, panitumumab, erlotinib, geftinib, and lapatinib
* Prior treatment with an EGFR inhibitor is allowed if it was administered as part of definitive therapy for locally advanced disease and completed >/=1 year before study enrollment
* Leptomeningeal disease as the only manifestation of the current malignancy
* Active infection requiring iv antibiotics
* Active autoimmune disease that is not controlled by non-steroidal anti-inflammatory drugs
* Current severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary, or metabolic disease; wound healing disorders; ulcers; bone fractures)
* History of heart failure or serious cardiac arrhythmia
* History of myocardial infarction within 6 months of Cycle 1, Day 1
* Clinically significant liver disease, including active viral, alcoholic or other hepatitis, cirrhosis, or current alcohol abuse
* HIV infection
* Primary central nervous system (CNS) malignancy or untreated/active CNS metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Pregnant or lactating women
* Malignancies other than SCCHN within 5 years prior to randomization, with the exception of adequately treated basal or squamous cell skin cancer and carcinoma in situ of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (tumor assessments according to RECIST criteria) | approximately 24 months

SECONDARY OUTCOMES:
Objective response: complete response or partial response | approximately 24 months
Disease control: complete response, partial response or stable disease | approximately 24 months
Duration of objective response | approximately 24 months
Time to disease progression | approximately 24 months
Overall survival | approximately 24 months
Safety: Incidence of adverse events | approximately 24 months
Pharmacokinetics: Cmax/Cmin | Pre-dose and 30 min after end of infusion on Day 1 of Cycles 1, 2, 3, and 4, and at treatment completion
Immunogenicity: anti-MEHD7945A levels | Pre-dose on Day 1 of Cycles 1 and 4, and at treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (47):
- United States (13):
  - Stanford, California
  - Aurora, Colorado
  - Miami, Florida
  - Chicago, Illinois
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Saint Joseph, Missouri
  - New York, New York
  - Chapel Hill, North Carolina
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Madison, Wisconsin
- Australia (6):
  - Darlinghurst, New South Wales
  - Waratah, New South Wales
  - Wollongong, New South Wales
  - Brisbane, Queensland
  - Kurralta Park, South Australia
  - Melbourne, Victoria
- Belgium (2):
  - Edegem
  - Namur
- Bulgaria (3):
  - Pleven
  - Rousse
  - Sofia
- France (3):
  - Clichy
  - Lyon
  - Villejuif
- Germany (2):
  - Berlin
  - Essen
- Hungary (3):
  - Debrecen
  - Győr
  - Szolnok
- Italy (4):
  - Udine, Friuli Venezia Giulia
  - Milan, Lombardy
  - Orbassano, Piedmont
  - Turin, Piedmont
- Romania (3):
  - Brasov
  - Cluj-Napoca
  - Timișoara
- Spain (4):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Salamanca, Salamanca
  - Valencia, Valencia
- United Kingdom (4):
  - Coventry
  - Glasgow
  - London
  - Sutton